CLINICAL TRIAL: NCT05150223
Title: The Effects of Functional Power Training on Attention, Gross and Fine Motor Skills, Participation and Quality of Life in Children With Attention Deficit Hyperactivity Disorder
Brief Title: The Effects of Functional Power Training in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-088
Record Dates: First submitted 2021-11-09; First posted 2021-12-09 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; Child Mental Disorder
Keywords: attention deficit; hyperactivity disorder; power; strength; training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional strength training group (Active Comparator): traditional strength training (running, jumping forward over a barrier with one leg and two legs, heel-rise, push up and ball throw with load, bench press, and flexion-abduction-external rotation pattern with theraband)
  Interventions: Other: traditional strength training
- Power Training group (Experimental): progressive functional strength training protocol (running, jumping forward over a barrier with one leg and two legs, heel-rise, push up and ball throw with load, bench press, and flexion-abduction-external rotation pattern with theraband)
  Interventions: Other: Power training
- Control group (No Intervention): no intervention Typically developing children

INTERVENTIONS:
Other: traditional strength training — traditional strength training (running, jumping forward over a barrier with one leg and two legs, heel-rise, push up and ball throw with load, bench press, and flexion-abduction-external rotation pattern with theraband). Participation in the traditional strength training group will complete these exercises with a load and without time limitations and speed.
  Arms: Traditional strength training group
Other: Power training — progressive functional strength training protocol (running, jumping forward over a barrier with one leg and two legs, heel-rise, push up and ball throw with load, bench press, and flexion-abduction-external rotation pattern with theraband)
  Arms: Power Training group

SUMMARY:
This study is aimed to investigate the effectiveness of functional power training on attention, gross and fine motor skill, participation and quality of life in children with attention deficit hyperactivity disorder (ADHD) by comparing traditional strength training and their healthy peers. In the literature, there are limited studies that investigate the effect of power exercise in children with ADHD. But there is no randomized controlled trial include power exercises which is designed to the National Strength and Conditioning Association (NSCA) criteria and investigate the effects on attention, gross and fine motor skill, participation and quality of life in children with ADHD. This study hypothesizes that power exercises could improve attention, gross and fine motor skill, participation, and quality of life better than traditional strength training in children with ADHD.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder is a neurodevelopmental disorder characterized by inattention, impulsivity, and hyperactivity. These core symptoms cause poor gross and fine motor skills. Recent critical review results suggest that motor performance not only consists of motor response activation. It also includes mental representation of activity, attention, memory, makes decisions, and control over preponderant responses. These findings support that ADHD symptoms could affect motor performance negatively. DSM-V (The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) also specifies the relationship between ADHD symptoms and poor motor performance. DSM-V pointed out motor difficulties that occur in ADHD are caused by inattention and impulsivity rather than neurological origin. In the literature, Tseng et al. investigated ADHD symptom's negative effect on motor performance in 42 school-aged children with ADHD. Tseng et al.'s study was shown that inattention and impulsivity were determinative symptoms for motor difficulties. Because of the ADHD's symptoms' effect on the motor skill, children with ADHD have poor fine manual control, manual coordination, body coordination, strength, and agility when they are compared with health peers.

These motor difficulties affect the academic, social, and daily life of children with ADHD. They have many restrictions on participation of daily living activities, school, social and sport activities and have decreased quality of life scores. It is considered that these symptoms of ADHD related to catecholamine systems. Jeyanthi et al. suggest that exercises both directly and indirectly affects catecholamine systems. In the literature, there are many studies that was included different exercise interventions involving children with ADHD. Many of the studies were shown that exercise had positive effects on ADHD symptoms. However, there is not enough information about the type, duration, intensity, and frequency of appropriate exercises. Power exercises can be an appropriate approach given the previously reported problems in children with ADHD. This type of exercise shown positive effects on the other populations (CP). The aim of the study is to investigate the effect of power exercises on children with ADHD by comparing these effects with traditional strength training and their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* • age between 6 years and 12 years;

  * Diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) by a child and adolescent health psychiatrist, regardless of subtype, according to DSM-V criteria
  * Have cognitive ability to follow instructions for assessment measures and exercise intervention

Exclusion Criteria:

* • Children have any other psychiatric diagnosis like autism spectrum disorder, psychotic symptoms, depression, etc.

  * Children have any neurological or orthopedic disorders like head injury, cerebral palsy, epileptic seizure, visual and speech disorder.

Inclusion Criteria for Healthy Children:

* Healthy children aged 6-12 years old
* Children without a psychiatric and neurological diagnosis

Exclusion Criteria for Healthy Children:

* Children got medical treatment for a neuropsychiatric disorder
* Children whose parents or themselves refused to participate

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Conners' Teacher Rating Scale (CTRS) | change from baseline to end of the 8 weeks
  CTRS is a reliable and valid 59-item teacher self-report form designed to identify children with ADHD and associated behavioral difficulties. Each item can be scored from 0 to 3; where 0 represents an item is not present and 3 represents an always or definitely present symptom.
Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) to measure motor proficiency. | change from baseline to end of the 8 weeks
  Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2) is norm referenced and designed to measure gross and fine motor skills in youth 4 to 21 years of age. Standard scores 40 are considered below average, whereas those >40 range from average to above average.
Evaluation of muscle power of lower extremity | change from baseline to end of the 8 weeks
  Muscle Power Sprint Test (MPST) will be used to assess lower extremity muscle power.Peak power and Mean Power (watts) were also calculated and used as markers of anaerobic power in the MPST. Power output for each sprint was calculated using body mass and running times, where power = (body mass Å~ distance2)/time. Peak power was defined as the highest calculated power, while Mean Power was defined as average power over the 6 runs.
Evaluation of muscle power of upper extremity | change from baseline to end of the 8 weeks
  Throw Basketball Test will be used to assess upper extremity muscle power. The distance from the starting line to where the ball landed was recorded in centimetres.

SECONDARY OUTCOMES:
The 30 seconds Repetition Maximum test | change from baseline to end of the 8 weeks
  The 30 seconds Repetition Maximum test was used to assess functional muscle strength of the lower extremities. The three closed kinetic chain exercises of lateral step-up test, Sit To Stand and attain stand through half knee were used. The children were instructed to perform as many repetitions as possible in 30 seconds for each of the exercises. Lateral step-up and attain stand through half knee were evaluated bilaterally. The repetition maximum for each side was used to calculate total scores for the left and right side and thus ﬁve ﬁnal scores were obtained.
walking speed | change from baseline to end of the 8 weeks
  1 Minute Walk Test (1 MWT) will be used to assess walking speed.
Evaluation of participation | change from baseline to end of the 8 weeks
  Participation and Environment Measurement Child & Youth (PEM-CY) is a parent-report questionnaire to assess participation and environment factors in the home, at school and within community Settings. The participation sections included 10 activities in the home setting, five activities in the school setting and 10 in the community setting. For each activity, parents are asked to determine the participation frequency (how frequently has the child participated with eight options: daily to never), participation involvement (how involved the child is while participating the activity rated on a five-point scale: very involved to minimally involved) and whether change is desired (do the parents want to see change in the child's participation in this type of activity: no or yes, with 5 different types of change).
Evaluation of quality of life | change from baseline to end of the 8 weeks
  The Pediatric Quality of Life Inventory (PEDS-QL) is a generic health related quality of life measure consisting of 4 core scales, physical function (8 items), emotional function (5 items), social function (5 items) and school function (5 items) that is intended for use in healthy and patient populations. Respondents are asked to recall the last month and indicate how frequently - from never to almost always - they have experienced specific phenomena. Item responses (0-100) are averaged to form total and core scores; higher scores indicate higher functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tseng MH, Henderson A, Chow SM, Yao G. Relationship between motor proficiency, attention, impulse, and activity in children with ADHD. Dev Med Child Neurol. 2004 Jun;46(6):381-8. doi: 10.1017/s0012162204000623. PMID 15174529
- [Background] S J, Arumugam N, Parasher RK. Effect of physical exercises on attention, motor skill and physical fitness in children with attention deficit hyperactivity disorder: a systematic review. Atten Defic Hyperact Disord. 2019 Jun;11(2):125-137. doi: 10.1007/s12402-018-0270-0. Epub 2018 Sep 27. PMID 30264226
- [Background] Cho H, Ji S, Chung S, Kim M, Joung YS. Motor function in school-aged children with attention-deficit/hyperactivity disorder in Korea. Psychiatry Investig. 2014 Jul;11(3):223-7. doi: 10.4306/pi.2014.11.3.223. Epub 2014 Jul 21. PMID 25110492
- [Background] Kaya Kara O, Livanelioglu A, Yardimci BN, Soylu AR. The Effects of Functional Progressive Strength and Power Training in Children With Unilateral Cerebral Palsy. Pediatr Phys Ther. 2019 Jul;31(3):286-295. doi: 10.1097/PEP.0000000000000628. PMID 31220015
- [Background] Moreau NG, Holthaus K, Marlow N. Differential adaptations of muscle architecture to high-velocity versus traditional strength training in cerebral palsy. Neurorehabil Neural Repair. 2013 May;27(4):325-34. doi: 10.1177/1545968312469834. Epub 2013 Jan 4. PMID 23292847
- [Background] Messler CF, Holmberg HC, Sperlich B. Multimodal Therapy Involving High-Intensity Interval Training Improves the Physical Fitness, Motor Skills, Social Behavior, and Quality of Life of Boys With ADHD: A Randomized Controlled Study. J Atten Disord. 2018 Jun;22(8):806-812. doi: 10.1177/1087054716636936. Epub 2016 Mar 24. PMID 27013028
- [Background] Goulardins JB, Marques JC, De Oliveira JA. Attention Deficit Hyperactivity Disorder and Motor Impairment. Percept Mot Skills. 2017 Apr;124(2):425-440. doi: 10.1177/0031512517690607. Epub 2017 Jan 31. PMID 28361657
- See also: National Strength and Conditioning Association — http://www.nsca.com/